CLINICAL TRIAL: NCT04912466
Title: A Phase 1a/1b Study Evaluating the Safety, Tolerability and Preliminary Efficacy of IBI322 Monotherapy or Combination Therapy in Subjects With Advanced Malignant Tumors.
Brief Title: IBI322 Monotherapy or Combination Therapy in Subjects With Advanced Malignant Tumors.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI322A105
Record Dates: First submitted 2021-05-28; First posted 2021-06-03 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IBI322 (Experimental): Singal arm
  Interventions: Drug: Biological: IBI322

INTERVENTIONS:
Drug: Biological: IBI322 — Recombinant anti-human CD47/PD-L1 bispecific antibody injection

SUMMARY:
The Phase Ia study was designed to evaluate the tolerability, safety, PK, PD, immunogenicity and primary resistance of single therapy tumor activity in subjects with advanced or metastatic solid tumors who have failed standard treatment. Phase Ib study was designed to evaluate the safety and initial efficacy of IBI322 in monotherapy or combination therapy in subjects with advanced or metastatic solid tumors. Investigators and sponsors determine the recommended dose of IBI322 for phase Ib based on PK, PD, safety and efficacy data obtained during phase Ia.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically/cytologically confirmed, locally advanced unresectable or metastatic tumors.
2. Per RECIST1, at least one evaluable or measurable lesion.
3. Male or female subject above 18 years old, no more than 75 years old.
4. Eastern Cooperative Oncology Group Performance Status (ECOG PS) performance status 0 or 1.
5. Must have adequate organ function

Exclusion Criteria:

1. Previous exposure to any anti-CD47 monoclonal antibody, SIRPα antibody, or CD47/SIRPα recombinant protein.
2. Direct coombs test was positive or have history of hemolytic anemia.
3. Subjects participating in another interventional clinical study, except for: observational (non-interventional) clinical studies or survival follow-up phase of interventional studies.
4. Patients who are on anticoagulants and /or require concomitant aspirin or other nonsteroids anti-inflammatory medications. Patients with a history of a bleeding diathesis (von Willebrand disease, end stage liver disease, hemophilia, etc.)
5. Subjects who have a history of blood transfusion within 2 weeks prior to the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2021-07-21 (Actual); Primary Completion 2022-12-03 (Actual); Study Completion 2023-08-25 (Actual)

PRIMARY OUTCOMES:
Number of DLT | 21 Days
Number of treatment related AEs | up to 90 days post last dose
Number of patients with response | Last patient enrolled+24 months

SECONDARY OUTCOMES:
Biomarker evaluation | from first dose until the date of first documented progression or date of death from any cause,whichever came first, assessed up to 24 months.
positive rate of ADA&NAB | from first dose until the date of first documented progression or date of death from any cause,whichever came first, assessed up to 24 months.
Area under the plsma concentration versus time curve(AUC) | Up to 90 days post last dose
Peak Plasma concentration(Cmax) | Up to 90 days post last dose
Clearance rate(CL) | Up to 90 days post last dose
the distribution volumn (Vd) | Up to 90 days post last dose
half-life period(t1/2) | Up to 90 days post last dose
Percentage of receptor occupancy | Up to 90 days post last dose
Hemoglobin level | Up to 90 days post last dose
Reticulocyte count (RET) | Up to 90 days post last dose
platelet count (PLT) | Up to 90 days post last dose

CONTACTS AND LOCATIONS:
Overall Officials: Jinming Yu, M.D., Principal Investigator — No.440, Jiyan Road, Jinang City, Shandong Province, China
Locations (1):
- Shandong Province Cancer Hospital, Jinan, Shandong, China